## Analytic plan Healthy Heart Habits (H^3)

NCT04158219

R03HL136540

3/8/22

## Analytic plan.

Means, standard deviations, frequencies, and percentages will be calculated to describe the sample. Because the intent of the open pilot trial was feasibility and acceptability assessment to inform additional treatment refinement, analysis will emphasize descriptive characterizations of the data and calculation of effect sizes to examine clinical magnitude of preliminary effects. Descriptive data on baseline characteristics and treatment engagement will be presented on the entire sample, regardless of trial completion. Treatment satisfaction and pre- to post- change were calculated only for completers. No correction for multiple comparisons will be made. Analyses were performed in Stata SE 16.